CLINICAL TRIAL: NCT00003066
Title: Phase II Evaluation of Docetaxel Combined With Estramustine Phosphate in Patients With Metastatic Breast Cancer
Brief Title: Docetaxel Combined With Estramustine in Treating Women With Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065737; CPMC-IRB-7929; NCI-V97-1325
Record Dates: First submitted 1999-11-01; First posted 2004-02-16 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2006-12

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Estramustine

INTERVENTIONS:
Drug: docetaxel
Drug: estramustine phosphate sodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of docetaxel combined with estramustine in treating women with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate, duration of response, duration of survival, and quality of life effects of docetaxel and estramustine combination in women with metastatic breast cancer.

OUTLINE: Patients receive estramustine 3 times a day for 3 days. Docetaxel begins on day 3 after the a.m. dose of estramustine and is given as a 1 hour infusion intravenously. Courses repeat every 21 days. If disease responds or is stable, treatment continues at the highest tolerance percentage of prescribed dose until appearance of disease progression. If complete response is documented, an additional 2 courses are given. Patients should receive a minimum of 2 courses unless rapid progression or unacceptable toxicity occur. Patients are followed monthly.

PROJECTED ACCRUAL: Approximately 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic breast cancer Measurable or evaluable disease Must be ineligible for other high priority national or institutional study No visible metastases on brain CT or MRI (unless single lesion amenable to surgical resection) Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: Over 18 Sex: Female Menopausal status: Not specified Performance status: ECOG 0-2 Life expectancy: More than 2 months Hematopoietic: WBC greater than 3,000/mm3 Platelet count greater than 100,000/mm3 No prior clotting disorder unless therapeutically anticoagulated Hepatic: Bilirubin less than the upper limit of normal SGOT or SGPT less than 1.5 times normal Renal: BUN less than 1.5 times normal Creatinine less than 1.5 times normal Cardiovascular: No prior thromboembolism unless therapeutically anticoagulated Other: No symptomatic ascites, pleural effusion or peripheral edema No serious medical or psychiatric illness No prior malignancy other than curatively treated carcinoma in situ of the cervix or skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy (2 weeks if weekly regimen) Any number of prior chemotherapy regimens allowed Endocrine therapy: Any number of prior hormonal therapy regimens allowed Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: At least 1 week since prior surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1997-02

CONTACTS AND LOCATIONS:
Overall Officials: Amy D. Tiersten, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center, New York, New York, United States